CLINICAL TRIAL: NCT03366870
Title: Efficacy of a Computerized Cognitive Behavioral Treatment for Insomnia: Increasing Access to Insomnia Treatment to Decrease Suicide Risk
Acronym: Vets Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Military Suicide Research Consortium (Other); Denver Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-0920
Record Dates: First submitted 2017-11-28; First posted 2017-12-08 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Insomnia; Physical Health Functioning; Mental Health Functioning
Keywords: CBT-I; Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computerized Intervention 1 (Experimental): A web-based program will deliver components of CBT-I on a time and event-based schedule. Pre and Post-Intervention assessments will be administered to determine the efficacy of the intervention.
  Interventions: Behavioral: Computerized Cognitive Behavioral Therapy for Insomnia
- Computerized Intervention 2 (Experimental): A web-based program will deliver components of sleep education via an Internet platform. Pre and Post-Intervention assessments will be administered to determine the efficacy of the intervention.
  Interventions: Behavioral: Sleep Education

INTERVENTIONS:
Behavioral: Computerized Cognitive Behavioral Therapy for Insomnia — A computerized insomnia intervention that employs the same behavioral, educational, and cognitive treatment components that underlie non-computerized CBT-I.
  Other Names: cCBT-I
  Arms: Computerized Intervention 1
Behavioral: Sleep Education — A web-based program will deliver components of sleep education via an Internet platform.
  Arms: Computerized Intervention 2

SUMMARY:
Insomnia is major problem among Operation Enduring Freedom (OEF), Operation Iraqi Freedom (OIF), and Operation New Dawn (OND) Veterans. Insomnia impacts physical and mental health functioning and is associated with reduced quality of life. Cognitive Behavioral Therapy for Insomnia (CBT-I) is one of the most promising treatments for insomnia; however, access to CBT-I is severely limited by a lack of trained clinicians within the Veterans Health Administration (VHA) and Department of Defense (DoD). There is a critical need to offer innovative approaches to meet the demand and need for insomnia treatment. Leveraging technology to meet treatment demands is consistent with service delivery models based upon stepped care principles. This randomized controlled trial will determine whether a computerized, self-guided, web-based version of CBT-I is efficacious in reducing insomnia symptoms and improving functioning compared to a computerized program control.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 55
2. History of deployment in the Global War on Terror
3. Eligible to receive care through VA ECHCS
4. Reliable access to the Internet
5. English speaking
6. Able to provide informed consent
7. Current insomnia diagnosis as defined by Diagnostic and Statistical Manual of Mental Disorders 5 (DSM 5) criteria

Exclusion Criteria:

1. Currently enrolled in/participating in other intervention research studies
2. Other untreated sleep disorders (e.g., sleep apnea, periodic limb movement)
3. Currently receiving formal psychological treatment for insomnia (not including sleep medications)
4. Past 3 month change in schedule and/or dosage of medications that are designed to improve/impact sleep
5. History of Bipolar Disorder (with manic episodes), Schizophrenia, Schizoaffective Disorder, or a Psychotic Disorder
6. Untreated seizures or seizure disorder
7. Physical illness that is active, unstable, degenerative, and/or progressive
8. Currently pregnant or plan to become pregnant in the next 6 months
9. Irregular work schedule, shift work, and/or life changes (e.g., new baby) interfering with regular sleep patterns
10. Significant cognitive impairment, as determined by chart review and/or during screening, that would interfere with ability to engage in SHUTi
11. Current non-alcohol Substance Use Disorder, excluding Cannabis Use Disorder, as determined by chart review and/or self-report screen of drug use (> 1 time) in past 3 months
12. Current Alcohol Use Diagnosis, as determined by SCID 5 module, in the past 3 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 250 (Actual)
Dates: Start 2018-03-24 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2020-06-16 (Actual)

PRIMARY OUTCOMES:
Change in Insomnia Symptom Severity as Measured by the Insomnia Severity Index | Baseline and 9 Weeks
  The primary analyses will be the intent-to-treat comparison between groups of the change in insomnia symptom severity as measured by the ISI from Time 1 to Time 2. Statistical inference regarding the difference between intervention groups will be based on the estimated coefficient for a group indicator variable in each of three analysis of covariance models with the change from Time 1 to Time 2 for each outcome serving as the dependent variable. Additional covariates will include the baseline value of the outcome to improve precision of the estimate, and any potential confounders discovered in the randomization check.
Maintenance of Change in Insomnia Symptom Severity as Measured by the Insomnia Severity Index at 6-months and 1-Year Post-Intervention | Baseline, 6-Months and 1-Year
  A similar analysis will be performed for the above noted insomnia severity outcome on the change from Time 1 to Time 3 and to Time 4 to determine persistence of group differences to six-months and one-year post-intervention.

SECONDARY OUTCOMES:
Change in Physical Health and Mental Health Functioning as Measured by the Veteran's SF-36 | Baseline and 9 Weeks
  A similar analysis will be performed with physical health and mental health functioning as the outcomes, based on self-reported responses to the Veteran's SF-36 measure.
Maintenance of Change in Physical Health and Mental Health Functioning as Measured by the Veteran's SF-36 at 6-months and 1-Year Post-Intervention | Baseline, 6-Months and 1-Year
  A similar analysis will be performed for the above noted outcomes on the change from Time 1 to Time 3 and to Time 4 to determine persistence of group differences to six-months and one-year post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Sarra Nazem, PhD, Principal Investigator — VHAECH
Locations (1):
- Rocky Mountain Regional VA Medical Center, Aurora, Colorado, United States

REFERENCES:
- [Derived] Nazem S, Barnes SM, Forster JE, Hostetter TA, Monteith LL, Kramer EB, Gaeddert LA, Brenner LA. Efficacy of an Internet-Delivered Intervention for Improving Insomnia Severity and Functioning in Veterans: Randomized Controlled Trial. JMIR Ment Health. 2023 Nov 24;10:e50516. doi: 10.2196/50516. PMID 37999953